CLINICAL TRIAL: NCT06162858
Title: Reaching Motion by the Elderly During Functional Activities. A Comparison Beween a Healthy Control Group and Patients With a Reverse Shoulder Arthroplasty
Brief Title: Reaching Motion During Functional Activities
Acronym: REACHRSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ONZ-2023-0416
Record Dates: First submitted 2023-11-06; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Shoulder Arthropathy Associated With Other Conditions; Healthy
MeSH Terms: interventions — 24,25-oxidolanosterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy participants (Other): no shoulder pain no shoulder diagnosis 60 years and older
  Interventions: Other: IMU (Inertial Measurement Devices)
- RSA participants (Other): primary reverse shoulder arthroplasty 60 years and older
  Interventions: Other: IMU (Inertial Measurement Devices)

INTERVENTIONS:
Other: IMU (Inertial Measurement Devices) — Functional placing and reaching of objects of different weights on different heights

SUMMARY:
Taking and moving objects is essential. When this becomes difficult, it affects daily functioning. This study aims to determine movement patterns, at the level of the shoulder, during different functional movements in elderly people aged 60 years and older. Movement patterns of people without shoulder problems and patients with a reverse shoulder prosthesis will be compared. These insights can contribute to improving functional rehabilitation in patients with a reverse shoulder prosthesis (RSA).

DETAILED DESCRIPTION:
This study aims to investigate how elderly people (60 years and older) without shoulder pain and patients with a reverse shoulder arthroplasty (60 years and older) perform functional reaching movements. Using IMUs (Inertial Measurement Units), the investigators want to look at mode of execution, relational positions of hand, elbow and shoulder in space, in relation to the trunk and each other, and any compensatory movements made by patients with a reverse shoulder arthroplasty.

At the time of testing, participants will first complete a series of questionnaires. These questionnaires will provide information about the daily functioning of all participants. The participants' shoulder strength will also be measured.

After applying the IMUs, the participant will first perform a maximal movement (active for participant) in 4 directions (forward and lateral lifting of arm, hand-to-neck , hand-to-back). Then the researcher will perform the same movements with the participant's arm (passive for participant). This will allow measurement of the maximum active and passive mobility of the shoulder. Next, the participant will be asked to place and take back a number of different objects (both in terms of size and weight) at predetermined heights.

The participants without shoulder pain will be tested once, the participants with a reverse shoulder arthroplasty we want to test 4 times. The participants without shoulder pain will be assigned to the control group. The participants with a reverse shoulder arthroplasty we want to test 4 times to monitor not only their movement pattern, but also any changes in this pattern .

The questionnaires, strength measurement and requested movements will be the same for both groups.

Analysis of these movements will provide us with insights that can help improve the functional rehabilitation of patients with a reverse shoulder prosthesis.

All participants with a reverse shoulder arthroplasty will be recruited at UZ, participants without shoulder pain will be recruited through different channels (these are not patients)

ELIGIBILITY:
Inclusion Criteria:

* 60 years and older
* no shoulder pain + no diagnosis of shoulder problem
* primary reverse shoulder arthroplasty

Exclusion Criteria:

* younger than 60 years
* shoulder pain at moment of testing
* known shoulder problem ( incl. diagnosis)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
IMU registration (3D kinematics upper limb) | healthy control group: baseline
  kinematic registration of performed exercises by all participants
IMU registration (3D kinematics upper limb) | RSA group: 3 weeks post surgery
  kinematic registration of performed exercises by all participants
IMU registration (3D kinematics upper limb) | RSA group: 6 weeks post surgery
  kinematic registration of performed exercises by all participants
IMU registration (3D kinematics upper limb) | RSA group: 12 weeks post surgery
  kinematic registration of performed exercises by all participants
IMU registration (3D kinematics upper limb) | RSA group: 6 months post surgery
  kinematic registration of performed exercises by all participants
IMU registration (3D kinematics upper limb) | RSA group: 12 months post surgery
  kinematic registration of performed exercises by all participants

SECONDARY OUTCOMES:
SPADI_DV | during procedure
  Content: 5 questions for the subscale pain and 8 questions for the disability subscale.
  Scoring: numeric rating scale from 1 to 10, with a maximum of 130. The total score is the sum of the sub-scores.
  Interpretation: The higher the score the more pain and disability. The lower the score, the better patients perceive their shoulder
Constant- Murley Score | during procedure
  Content: partially clinical (65 points) and partially PROM (35 points) assessed.
  Scoring: The formula to calculate the total score is:" pain (0-15) + ADL (4x (0-5) = 0-20) + mobility (4 x (0-10) = 0-40)
  + strength (0 -25)". Strength will be measured with the arm elevated to 90 ° in the scapular plane using an IDOmeter.
  Interpretation: 0-55 points = bad, 56-70 points = mediocre, 71-85 points = good, 86-100 points = excellent score
EQ5D5L | during procedure
  Content: 5 questions + EQ-5D VAS for general health. Scoring: 5-response scale (from 'no problems' to 'extreme problems') + VAS percentage between 0 (worst imaginable health state) and 100 (best imaginable health state).
  Interpretation: VAS score for general health indicates how a patient perceives his general health, Other questions are descriptive for problems in mobility, self-care, usual activities, pain/ discomfort, anxiety/depression
VAS-pain | during procedure
  Pain is scored between 0 and 10. 0 = no pain, 10= worst possible pain
AROM | during procedure
  active range of motion for forward flexion, abduction, hand-to-neck, hand-to-back forward flexion and abduction with extended elbow, functional internal and external rotation in standing position.
  * maximal pain free ROM
  * forward flexion and abduction with extended elbow: measured with the EasyAngle (Meloq AB Sweden)
  * hand-to-back and hand-to-neck test : scored as in Constant-Murley Score
PROM | during procedure
  passive range of motion for forward flexion and abduction
  * maximal pain free ROM
  * measured with the EasyAngle (Meloq AB Sweden)
strength | during procedure
  strength will be measured for forward flexion in 0° elevation and in 90° elevation with the EasyForce.
  FF at 0° elevation: participants will sit on a chair without backrest, both feet on the ground. Arm in neutral rotation, hand in a fist, thumb facing upward FF at 90° elevation: participants will stand, the arm with extended elbow held at 90° elevation (FF). Hand in a fist, thumb facing upward

OTHER OUTCOMES:
AGE | during procedure
  specify age of participant
GENDER | during procedure
  specify age of participant
DOMINANCE | during procedure
  specify hand dominance of participant
height | during procedure
  specify participants height
weight | during procedure
  specify participants weight

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Van Tongel, PhD, Principal Investigator — University Hospital Ghent, University Ghent; Ann Cools, PhD, Study Chair — University Ghent; Annelies Maenhout, PhD, Study Chair — University Ghent
Locations (2):
- Belgium (2):
  - Ghent University Hospital, Ghent
  - University Ghent, Ghent

IPD SHARING:
Plan to Share IPD: No